CLINICAL TRIAL: NCT04787523
Title: Rectrospect - a Study on the Immun Cell Infiltrate in a Retrospective Rectal Cancer Cohort.
Brief Title: Rectrospect - a Retrospective Study of Treatment Response
Acronym: Rectrospect
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Angenete, Professor, Sahlgrenska University Hospital
Other Study IDs: Rectrospect
Record Dates: First submitted 2021-02-27; First posted 2021-03-08 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biopsies taken at diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pathological response to treatment: Response evaluated using the pathology report
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Patients have received neoadjuvant radiotherapy

SUMMARY:
Biopisies from patients diagnosed with rectal cancer between 2007-2019 will be cut into 4-6 micrometer thin sections for morphology and immunostaining. Every section will be numbered with a code that is connected to the patients personal identification number and the code list will be kept separately from the biopsies in a password protected file on the Sahlgrenska University Hospital server.

Patient data and outcome regarding response to treatment will be collected from patient charts and the Swedish ColoRectal Cancer Registry, but all data will be numbered with the same code number and all results will be kept away from the code list. In order to achieve the stated aims, that is, to study how the molecular and cellular characteristics of the tumour and its surrounding microenvironment as well as the interaction of tumour cells and immune cells affect treatment response, several molecular and cellular techniques and assays may be applied.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer and treatment between 2007 and 2019

Exclusion Criteria:

* No rectal cancer or no neoadjuvant treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with neoadjuvant treatment between 2007-2019
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Immun cell infiltrate in pathology sections from the tumour | Biopsies taken preoperatively
  Number of of CD3+ and CD8+ cells in the tumour in relation to response to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No